CLINICAL TRIAL: NCT01430806
Title: Dronedarone for Patients With Recurrent ICD Shocks Due to Ventricular Arrhythmia Resistant to Their Antiarrhythmic Drug Therapy or Ablation
Brief Title: Dronaderone to Prevent Recurrent Implantable Cardioverter Defibrillator (ICD) Shocks
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, moti haim, Director, Electrophysiology Service,, Rabin Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6402
Record Dates: First submitted 2011-09-07; First posted 2011-09-08 (Estimated); Last update posted 2011-09-08 (Estimated); Status verified 2011-09

CONDITIONS: ICD; ICD SHOCKS; DRONEDARONE
MeSH Terms: interventions — Dronedarone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dronedrone Arm (Other)
  Interventions: Drug: Dronedarone arm; Drug: Dronedarone

INTERVENTIONS:
Drug: Dronedarone arm — PO Dronedarone 400 mg BID
Drug: Dronedarone — Dronedarone PO 400 MG BID

SUMMARY:
Recurrent ICD shocks are a serious problem in pts with ICD. Treatment failure with other antiarrhythmics and ablation are common. Dronedarone is a new antiarrhythmic drug with ion channel properties similar to amiodarone.

Several case reports have shown promising results with Dronedarone for this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Recurernt ICD shocks depite other antiarrhythmic drug therapy

Exclusion Criteria:

* CHF NYHA IV OR DECMPENSATED III
* PERMANENT AF
* LIVER DYSFUNCION
* CR CLEARANCE <30

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-10; Primary Completion 2014-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Number of ICD shocks due to VT in the 6 months period after starting Dronedarone | 1 year